CLINICAL TRIAL: NCT00652262
Title: An Open, Multi-centre, Flexible Dose Uptitration Study to Investigate the Efficacy and Safety of Vardenafil 10 mg and 20 mg in Males With Spinal Cord Injury Suffering From Erectile Dysfunction
Brief Title: BAY38-9456 - Supportive Trial for Spinal Injury
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 100608
Record Dates: First submitted 2008-04-01; First posted 2008-04-03 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Erectile Dysfunction; Sexual Dysfunction; Spinal Cord Injury
Keywords: Vardenafil; PDE5 inhibitor; Erectile dysfunction; Spinal cord injury
MeSH Terms: conditions — Erectile Dysfunction; Sexual Dysfunction, Physiological; Spinal Cord Injuries | interventions — Vardenafil Dihydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Levitra (Vardenafil, BAY38-9456)

INTERVENTIONS:
Drug: Levitra (Vardenafil, BAY38-9456) — Patients received BAY 38-9456 10 mg for the first 4 weeks of the treatment period, and then went on to receive 10 mg or 20 mg for the following 8 weeks.

SUMMARY:
BAY 38-9456 10 mg and 20 mg can be given as safe and efficacious medications to patients with spinal cord injury suffering from erectile dysfunction, and that erectile dysfunction can be improved by uptitration to BAY 38-9456 20 mg when the treatment with 10 mg is not sufficiently effective

ELIGIBILITY:
Inclusion Criteria:

* Male with erectile dysfunction according to the NIH Consensus Statement (inability to attain and/or maintain penile erection sufficient for satisfactory sexual performance), solely as a result of a traumatic injury to the spinal cord (suffering more than 6 months ago)
* Patients answering "yes" to the question regarding the presence of residual erectile function over the past 6 months [At home over the past 6 months, have you experienced at least some enlargement of your penis in response to: (1) mechanical stimulation by yourself or your partner, or (2) visual stimulation?]

Exclusion Criteria:

* History of diabetes mellitus
* Patients who are taking nitrates or nitric oxide donors
* Patients who have experienced no enlargement of penis with PDE5 inhibitor and/or who have withdrew the use of PDE5 inhibitor due to ADRs

Ages: 20 Years to 64 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2004-03; Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
The Erectile Function (EF) domain score of IIEF calculated as the sum of scores from Questions 1 to 5 and 15 | At 12 weeks after start of study drug administration using data at LOCF to account for dropouts

SECONDARY OUTCOMES:
The Global Assessment Question | At 4, 8, 12 weeks after start of study drug administration and LOCF
The IIEF EF domain score | At 4, 8, 12 weeks after start of study drug administration
IIEF domain scores other than the EF domain score[intercourse satisfaction (Q6 to Q8), overall satisfaction (Q13, Q14), orgasmic function (Q9, Q10), sexual desire (Q11, Q12)] | At 4, 8, 12 weeks after start of study drug administration and LOCF
Scores of Questions 1 to 15 on the IIEF Questionnaire | At 4, 8, 12 weeks after start of study drug administration and LOCF
Patient's diary response concerning hardness of erection, maintenance of erection, satisfaction with overall hardness of erection, ability of insertion, overall satisfaction with sexual experience and ejaculation | At 4, 8, 12 weeks after start of study drug administration and LOCF
Safety data | Throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (3):
- Japan (3):
  - Nagoya, Aichi-ken
  - Iizuka, Fukuoka
  - Beppu, Oita Prefecture